CLINICAL TRIAL: NCT05906134
Title: A Randomized Controlled Trial Comparing Local Intercostal Nerve Blocks, Cryo-ablation Plus Intercostal Nerve Blocks, and Serratus Plane Catheter Plus Intercostal Nerve Blocks After Minimally Invasive Esophagectomy
Brief Title: Minimally Invasive Esophagectomy Pain Control Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rib Block 21181
Record Dates: First submitted 2023-01-30; First posted 2023-06-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain, Acute; Postoperative Complications
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: The randomization method will be sealed opaque envelopes with computer generated numbers inside that will have been created at the start of the study. The envelopes will be kept in the Thoracic Surgery clinic by the research coordinator. At the time of randomization, the envelope will be picked from random for each patient designating which group they will be assigned to. The anesthesia team, the thoracic surgeon performing the surgery, and the thoracic surgery clinical fellows for the study will be made aware of what arm the subject is part of for preoperative planning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- local intercostal nerve block (Active Comparator): Patients receiving intercostal blocks will receive a total of 1.0 cc/kg of 0.25% Bupivacaine + epinephrine. This will be divided into two-thirds allocated for use in the chest/intercostal block and one-third allocated for use in the abdomen.
  Interventions: Procedure: Local intercostal nerve block; Procedure: Thoracic epidural catheter
- cryo-ablation plus intercostal nerve block (Active Comparator): Patients receiving cryo-analgesia and intercostal blocks, the patient will receive cryo-ablation prior to the intercostal block. The cryo-ablation will occur 2 cm from the sympathetic chain 2 intercostal spaces above and 2 intercostal spaces below the access incision. The patient will also receive a total of 1.0 cc/kg of 0.25% Bupivacaine + epinephrine. This will be divided into two-thirds allocated for use in the chest/intercostal block and one-third allocated for use in the abdomen.
  Interventions: Procedure: Cryo-analgesia and intercostal nerve block; Procedure: Thoracic epidural catheter
- serratus plane catheter plus intercostal nerve block (Active Comparator): Patients receiving serratus plane catheter blocks and intercostal nerve blocks, a total of 1.0 cc/kg of 0.25% Bupivacaine + epinephrine will be administered. A total of 20 cc of the weight-based calculation will be reserved for the serratus plane catheter. The remaining local anesthetic will be divided into two-thirds for the chest and one-third for the abdomen. Patients with serratus plane catheters will have an ongoing infusion of 0.2% ropivacaine at 8 ml per hour. The serratus plane catheters will also receive a bolus of 20 ml of 0.25% bupivacaine with epinephrine on Post Operative Day (POD) #1, 2, 3, 4, and 5 by the pain service.
  Interventions: Procedure: Serratus plane catheter blocks and intercostal nerve blocks; Procedure: Thoracic epidural catheter

INTERVENTIONS:
Procedure: Local intercostal nerve block — Patients receiving intercostal blocks will receive a total of 1.0 cc/kg of 0.25% Bupivacaine + epinephrine. This will be divided into two-thirds allocated for use in the chest/intercostal block and one-third allocated for use in the abdomen.
  Arms: local intercostal nerve block
Procedure: Cryo-analgesia and intercostal nerve block — The cryo-ablation will occur 2 cm from the sympathetic chain 2 intercostal spaces above and 2 intercostal spaces below the access incision. The patient will also receive a total of 1.2 cc/kg of 0.25% Bupivacaine + epinephrine. This will be divided into two-thirds allocated for use in the chest/intercostal block and one-third allocated for use in the abdomen.
  Other Names: Cryo-ablation
  Arms: cryo-ablation plus intercostal nerve block
Procedure: Serratus plane catheter blocks and intercostal nerve blocks — A total of 1.2 cc/kg of 0.25% Bupivacaine + epinephrine will be administered. A total of 20 cc of the weight-based calculation will be reserved for the serratus plane catheter. The remaining local anesthetic will be divided into two-thirds for the chest and one-third for the abdomen. Patients with serratus plane catheters will have an ongoing infusion of 0.2% ropivacaine at 8 ml per hour. The serratus plane catheters will also receive a bolus of 20 ml of 0.25% bupivacaine with epinephrine on POD #1, 2, 3, 4, and 5 by the pain service.
  Arms: serratus plane catheter plus intercostal nerve block
Procedure: Thoracic epidural catheter — The pain service and thoracic surgery attending physician will assess if the patient's pain is not well-controlled using the pain modality they are randomized to. If additional pain control is needed, this will likely consist of a thoracic epidural catheter.
  Any additional pain control will be added as an adjunct to the study arm and will be noted in the data set.

SUMMARY:
A pilot randomized controlled trial comparing intercostal nerve blocks, cryo-ablation plus intercostal nerve blocks, and serratus plane catheter plus intercostal nerve blocks in patients undergoing esophagectomies with minimally invasive thoracic approaches.

DETAILED DESCRIPTION:
Pilot study planned to consent 30 patients in total with a projected study timeline of 2-3 years for completion. Participants will be enrolled in the study and randomized in their preoperative clinic visit. On the day of surgery, they will receive the intervention they were randomized to. 10 patients will be randomized to the intercostal block group, 10 patients will be randomized to the cryo-ablation plus intercostal block group, and 10 patients will be randomized to the serratus plane catheter plus intercostal block group. They will be followed throughout their hospital stay until discharge for data collection purposes. Once the patient is discharged from the hospital, post-operative follow-up in the Swedish Thoracic Surgery Clinic will be collected up to 1 year post-operatively.

ELIGIBILITY:
Inclusion Criteria:

All adult individuals who undergo an esophagectomy with an intended minimally invasive approach of the chest at Swedish Medical Center-First Hill. These approaches include:

* 3-hole with R video-assisted thoracoscopic surgery (VATS)
* Ivor Lewis R VATS

Exclusion Criteria:

* Age <18
* Unable to consent
* Additional surgical procedures planned
* Patients with previous thoracic surgery
* Patient with chronic pain on a daily regimen of narcotics
* Non-English speaking
* Contraindications to neuraxial anesthesia (ongoing anticoagulation, anticipated post-operative therapeutic anticoagulation, spinal cord stimulators, anatomic abnormalities preventing epidural placement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pain Change Over Time | Baseline (prior to OR) to every 12 hours postoperatively thru Post Operative Day 4.
  Compare post-operative pain score changes over time between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain | Baseline (Prior to OR)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain | Post-Op Time 0
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 1 (AM) | Post Operative Day 1 (AM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 1 (PM) | Post Operative Day 1 (PM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 2 (AM) | Post Operative Day 2 (AM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 2 (PM) | Post Operative Day 2 (PM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 3 (AM) | Post Operative Day 3 (AM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 3 (PM) | Post Operative Day 3 (PM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 4 (AM) | Post Operative Day 4 (AM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.
Post Operative Pain Day 4 (PM) | Post Operative Day 4 (PM)
  Compare single timepoint post-operative pain scores between intercostal nerve blocks, cryo-analgesia, and serratus plane catheters in patients undergoing minimally invasive esophagectomy. Patients will be asked specifically about thoracic/chest pain and asked to rate this pain on a Likert pain scale of 0-10, 0 being no pain and 10 being the worst pain they can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Louie, M.D., Principal Investigator — Swedish Cancer Institute
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States